CLINICAL TRIAL: NCT01524523
Title: Biochemical and Genetic Mechanisms of Acute Clinical Pain During Bone Marrow Aspiration
Brief Title: Bone Marrow Aspiration Pain Study
Status: Withdrawn | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120001; 12-CC-0001
Record Dates: First submitted 2012-02-01; First posted 2012-02-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2013-06-27

CONDITIONS: Acute Pain; Gene Expression; Nitric Oxide
Keywords: Gene Expression; Acute Pain; Nitric Oxide; Pain; Bone Marrow
MeSH Terms: conditions — Acute Pain; Pain

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Many people feel pain during and after bone marrow aspiration (collection). Studies suggest that pain may be related to different kinds of inflammation, or the presence of nitric oxide (a normally occurring gas) in the body. Researchers want to study nitric oxide levels in the blood and breath before and after bone marrow collection. They will look at how these levels relate to feelings of pain.

Objectives:

- To better understand pain related to having a bone marrow collection.

Eligibility:

- Individuals at least 18 years of age who are enrolled in a study that requires bone marrow collection.

Design:

* Participants will be screened with a physical exam, medical history, and blood sample.
* Participants will provide study blood and breath samples to check nitric oxide levels. Participants will also have a test to measure skin sensitivity to heat and touch.
* During the collection, participants will keep track of their pain levels.
* After the collection, participants will keep track of any pain medications they take. They will also record if and when they eat any foods that contain nitrates for about 24 hours.

DETAILED DESCRIPTION:
Abstract:

This project will explore the biochemical mechanisms associated with acute pain produced by bone marrow aspiration in 36 healthy subjects by : 1) Evaluation of any strong relationships of NO metabolism (as measured by plasma nitrite, nitrosated proteins, cyclic GMP, plasma hemoglobin, reticulocytes, as well as markers of inflammation) with the levels of acute pain in healthy subjects and; 2) Identification of differentially expressed genes and proteins as markers for the nature and severity of pain from bone marrow aspiration. Elucidation of these relationships may identify novel targets for intervention leading to attenuation of pain, improved treatment and less impact on quality of life (QOL) and may identify potential mechanisms for the role of NO in other inflammatory or pain syndromes.

Objectives:

The first objective of the study is to characterize genetic expression during acute pain and pain free phases pre and post bone marrow aspiration (BMA). The second objective is to measure at multiple time points levels of exhaled Nitric Oxide (eNO) and other biomarkers in subjects during pre- and post BMA. The third objective is to evaluate acute and experimental pain perception in these subjects.

Population:

This study will recruit healthy subjects (N=36) who have agreed to donate bone marrow.

Design:

This is a prospective, exploratory study of sensory and affective pain in healthy volunteers. Participants will undergo evaluations (eNO, blood collection, and quantitative sensory testing) during a clinic visit to undergo bone marrow aspiration.

Importance:

The purpose of this study is to improve the understanding of the biochemical and molecular genetic mechanisms associated with acute pain in a healthy population by characterizing the leukocyte transcriptome of pain pre- and post BMA. It is hypothesized that analysis of the transcriptome will result in a panel of biomarkers that correlate with acute pain in a healthy population. The successful elucidation of these relationships may identify novel targets for intervention leading to attenuation of pain, improved treatment and less impact on quality of life and functional status.

ELIGIBILITY:
* INCLUSION CRITERIA FOR SUBJECTS:

All subjects enrolled in the parent protocol are eligible for enrollment in this study provided they have met all the inclusion criteria in the parent protocol and if they meet all of the following criteria:

* Age greater than or equal to 18 years old.
* No chronic medication use that in the judgment of the investigators could confound the study or biomarker measurements.
* Can speak and understand English to complete assessments and scales

EXCLUSION CRITERIA FOR ALL STUDY PARTICIPANTS:

Study participants will be excluded from the study if he/she has one or more of the following:

* Inability to provide informed consent.
* Drug or alcohol dependence/abuse within the past 5 years
* Cigarette smoking or the use of any tobacco products within two years
* Use of tranquilizers, steroids, and non-steroidal anti-inflammatory agents three or more times per week.
* Clinically significant medical condition that will confound the analysis of factors associated with pain, such as:

  * Chronic inflammatory disease (i.e. rheumatoid arthritis, systemic lupus erythematosus, cirrhosis)
  * Chronic pain condition
  * Diabetes mellitus
  * Known malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12-02; Study Completion 2013-06-27

PRIMARY OUTCOMES:
Differences over time between whole blood gene expression in the peripheral blood of healthy subjects undergoing an acute pain stimulus.

SECONDARY OUTCOMES:
Quantification and differences in laboratory correlates (particularly plasma nitrite, nitrosated proteins, and cyclic GMP) in health subjects pre- and post-BMA.
Quantification of pain sensory perception in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Wendy B Smith, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)

REFERENCES:
- [Background] Vichinsky EP, Styles LA, Colangelo LH, Wright EC, Castro O, Nickerson B. Acute chest syndrome in sickle cell disease: clinical presentation and course. Cooperative Study of Sickle Cell Disease. Blood. 1997 Mar 1;89(5):1787-92. PMID 9057664
- [Background] The labrets of the northern "Esquimaux" (1826). Alaska Med. 1991 Apr-Jun;33(2):93. No abstract available. PMID 1892235
- [Background] McKerrell TD, Cohen HW, Billett HH. The older sickle cell patient. Am J Hematol. 2004 Jun;76(2):101-6. doi: 10.1002/ajh.20075. PMID 15164373